CLINICAL TRIAL: NCT02003729
Title: SIESTA: Home Sleep Study With ApneaDx™ for the Diagnosis of Obstructive Sleep Apnea: A Pragmatic Randomized Controlled Trial
Brief Title: SIESTA: Home Sleep Study With ApneaDx™ for the Diagnosis of Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: Mars, Inc. (Industry)
Responsible Party: Principal Investigator, Murray Krahn, MD, MSc, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 29539
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; Portable Monitor; AHI; ESS; Cost effectiveness
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Portable Sleep Monitor (Active Comparator): The clinical diagnosis of OSA will be done according to the American Academy of Sleep Medicine criteria, a combination of data from clinical examination, presenting symptoms, risk factors and results from portable monitor sleep studies.
  Interventions: Device: Portable Sleep Monitor
- Polysomnography (No Intervention): The clinical diagnosis of OSA will be done according to the American Academy of Sleep Medicine criteria, a combination of data from clinical examination, presenting symptoms, risk factors and results from polysomnography from the sleep clinic.

INTERVENTIONS:
Device: Portable Sleep Monitor — ApneaDx™ is a new PM that uses a microphone to record breath sounds and an acoustical analysis algorithm of breath sounds to determine the AHI.
  Other Names: ApneaDx
  Arms: Portable Sleep Monitor

SUMMARY:
The SIESTA Home Sleep Study is a pragmatic, multi-centre randomized single-blinded two arm trial, assisted by a Decision Analytic Model, primarily designed to assess the accuracy, effectiveness and cost-effectiveness of diagnosing OSA assisted by ApneaDx™ as compared to PSG as a reference standard.

DETAILED DESCRIPTION:
In Ontario, approximately 130,000 sleep studies were conducted in 2008, which is twice the number of sleep studies reported in 1999. In 2008, Ontario spent approximately $40 million on polysomnography (PSG) testing alone, despite the fact that access to PSG remained limited, with an average waiting time of approximately 3.5 months for an in-laboratory sleep study and approximately 12 months from referral to appropriate treatment. Portable monitors (PM) have been developed in an effort to substitute for the more costly and labor intensive clinic-based PSG. As of 2011, there are over 40 PM commercially available in the United States with different configurations for cardiorespiratory and neurophysiologic signals.

At the request of the Ontario Health Technology Advisory Committee (OHTAC), a panel that makes recommendations to the Ontario Ministry of Health and Long-Term Care about the uptake and diffusion of health technologies, the Toronto Rehabilitation Institute convened an expert panel in 2007 to explore alternative approaches to the diagnosis of obstructive sleep apnea (OSA). Members of the expert panel suggested that despite the availability of a large number of PMs, home assessments are problematic as technicians are required to ensure continuous placement of electrodes for reliable testing. They also suggested that a good screening tool was not available at that time. The Toronto Rehabilitation Institute therefore undertook a research study that eventually led to the development of the ApneaDx™ PM.

ApneaDx™ is a new PM that uses a microphone to record breath sounds and an acoustical analysis algorithm of breath sounds to determine the (Apnea Hypopnea Index) AHI. Results from preliminary studies suggest that the AHI derived from ApneaDx™ approximates that from PSG. In preliminary studies, it appears that for the diagnosis of sleep apnea, home sleep study with ApneaDx™ is simple and reliable even when conducted by untrained users.

This study evaluates the effectiveness and cost-effectiveness of OSA diagnosed assisted by a home sleep study with ApneaDx™. This study will be conducted by the Toronto Health Economics and Technology Assessment (THETA) Collaborative. Data from this study will be used to support practice recommendations regarding the use of a home sleep study with ApneaDx™ as input for diagnosis of OSA by the OHTAC and reimbursement considerations by the Ontario Ministry of Health and Long-Term Care.

ELIGIBILITY:
Inclusion Criteria:

* Referral to a sleep clinic by a general practitioner or family physician with symptoms suggestive of OSA.
* Provide signed informed consent
* At least 18 years of age
* Ability to complete study questionnaires either on their own or with assistance

Exclusion Criteria:

* An existing diagnosis of other sleep disorders (eg, periodic limb movement disorder);
* A history of neuromuscular diseases (e.g., multiple sclerosis, muscular dystrophy)
* A history of congestive heart failure
* A history of stroke/Transient Ischemic Attack
* a history of chronic respiratory diseases (e.g., asthma, chronic obstructive pulmonary disease, lung cancer, cystic fibrosis and occupational lung diseases)
* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the accuracy of the clinical diagnosis of OSA | 4-5 months
  • To evaluate the accuracy of the clinical diagnosis of OSA assisted by the home sleep study with ApneaDx against the clinical diagnosis assisted by the in-laboratory sleep study, PSG as the reference standard.
To evaluate the agreement between the Apnea Hypopnea Index (AHI) from the home sleep study with ApneaDx™ and the in-laboratory sleep study with polysomnography (PSG) | 5 months
  • To evaluate the agreement between the AHI from the home sleep study with ApneaDx™ and the in-laboratory sleep study with PSG in patients being referred to sleep clinics with suggestive OSA symptoms.

SECONDARY OUTCOMES:
To evaluate the cost-effectiveness (cost per quality-adjusted life year) of the OSA | 4-5 months
  • To evaluate the cost-effectiveness (cost per quality-adjusted life year) of the OSA after diagnosis based on home sleep study with ApneaDx™ in comparison with after diagnosis based on an in-laboratory sleep study with PSG.

CONTACTS AND LOCATIONS:
Overall Officials: Murray Krahn, MSc, MD, Principal Investigator — University of Toronto
Locations (1):
- Sleep Disorders Laboratory, Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Fitzpatrick M, Rac VE, Mitsakakis N, Abrahamyan L, Pechlivanoglou P, Chung S, Carcone SM, Pham B, Kendzerska T, Zwarenstein M, Gottschalk R, George C, Kashgari A, Krahn M. SIESTA - Home sleep study with BresoDx for obstructive sleep apnea: a randomized controlled trial. Sleep Med. 2020 Jan;65:45-53. doi: 10.1016/j.sleep.2019.07.013. Epub 2019 Jul 22. PMID 31707288